CLINICAL TRIAL: NCT01759693
Title: Platelet Activation in Chronic Inflammatory Skin Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0113; MMC 0113 (Other: Meir Medical Center)
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Urticaria; Atopic Dermatitis
Keywords: Platelet activation
MeSH Terms: conditions — Urticaria; Dermatitis, Atopic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Skin disease: Patients with urticaria or atopic dermatitis
  Interventions: Procedure: Blood sampling
- Control: Healthy volunteers
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling

SUMMARY:
Platelets are blood cells that are important in coagulation of the blood. These cells have recently been shown to play a role in a number of other biologic processes, for example inflammation. In this study the investigators will determine the extent of platelet activation in people suffering from common chronic skin inflammation-urticaria and allergic dermatitis.

ELIGIBILITY:
Inclusion Criteria: Urticaria or atopic dermatitis -

Exclusion Criteria:Lack of informed consent

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Platelet activation | 6 months
  Platelet function will be assessed at enrollment

SECONDARY OUTCOMES:
Mean platelet volume | 6 months
  Mean platelet volume will be assessed at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel